CLINICAL TRIAL: NCT04829643
Title: Targeting the Future of Axillary Staging in Early Breast Cancer: A Comparative Study: Sentinel Node Biopsy vs PET/MRI
Brief Title: Axillary Staging in Early Breast Cancer: SNB vs PET/MRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Collaborators: IBFM- Consiglio Nazionale delle Ricerche (Unknown)
Responsible Party: Principal Investigator, Oreste Davide Gentilini, Head of Breast Unit, Head of Breast Surgery, IRCCS San Raffaele
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SNBvsPET/MRI 2
Record Dates: First submitted 2021-03-31; First posted 2021-04-02 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2024-10

CONDITIONS: Breast Cancer; Sentinel Lymph Node; Early-stage Breast Cancer
Keywords: PET/MRI; sentinel node biopsy; early breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PET/MRI (Experimental): Patients with early breast cancer up to 3 cm without overt nodal involvement who are candidates to upfront surgery
  Interventions: Diagnostic Test: PET/MRI

INTERVENTIONS:
Diagnostic Test: PET/MRI — A consecutive cohort of 247 patients with early BC and no suspicious nodes at both clinical and A-US evaluations and candidates to upfront surgery and SNB will be recruited

SUMMARY:
The gold standard of surgical treatment for patients with early breast cancer (BC) is breast conservation and sentinel node biopsy (SNB). Ongoing randomized trials are evaluating to omit surgery at all when axillary imaging is negative. However, the available diagnostic tools still have several limitations in accuracy.

Combining the specificity of PET, with the superior sensitivity of MRI, hybrid PET/MRI might be a non-invasive, one-stage, operator-independent imaging method to accurately define nodal status and, whenever negative, might replace surgery for axillary staging.

The project includes patients with <3 cm BC without overt nodal involvement who will undergo PET/MRI prior to surgery. The primary aim is to compare the staging power between SNB and PET/MRI in detecting axillary lymph node macrometastases (>2 mm). Additionally, general concordance and diagnostic accuracy of PET/MRI vs SNB, eventual correlation with BC molecular subtypes and MRI findings will be evaluated.

DETAILED DESCRIPTION:
SNB is the gold standard for axillary staging in early BC patients. Although being a minimally invasive, it is time consuming both for surgeon and pathologist, it may add a further scar and is not free from complications: seroma, limitation of shoulder movement, nerve injury, lymphedema. To date, patients undergoing breast conserving surgery (BCS) with 1 to 2 positive nodes can be treated with SNB alone (ACOSOG Z011 trial NCT00003855[2-4]) and researchers are evaluating within large randomized trials to even omit surgery at all when axillary imaging is negative (SOUND (Sentinel node biopsy vs Observation after axillary Ultra-souND), PI and Study Chair Dr.O.Gentilini,MD, NCT02167490 and INSEMA (Intergroup-SEntinel-MAmma) trial NCT02466737.

While the role of surgery is decreasing, the role of preoperative imaging is increasing. In the future, imaging might even replace surgery in the axillary staging of BC patients, still providing an appropriate level of information to guide medical treatments which are more and more tailored on biology rather than on nodal status. In this context, an unmet need is to achieve the most accurate preoperative imaging assessment of the axilla in order to decide the appropriate treatment for each patient.

The hypothesis of this project is that PET/MRI might provide a single, one-stage, non-invasive, operator independent imaging modality in patients with small BC allowing to select the proper treatment for patients. PET/MRI is a relatively new imaging tool and its field of application is still object of scientific speculation.

ELIGIBILITY:
Inclusion Criteria:

* signed Informed Consent
* age > 18
* non palpable lymph nodes
* no suspicious nodes at A-US (Axillary- ultrasound)
* candidate to mastectomy or breast conserving surgery and BLS (Sentinel Node Biopsy)

Exclusion Criteria:

* pregnancy
* distant metastasis
* inflammatory cancer
* claustrophobia
* allergy to contrast agent
* severe renal insufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
SNB vs PET/MRI | Within 1 month after surgery
  Results from SNB will be compared to results from PET/MRI y results from SNB will be available and compared to results of preoperative PET/MRI

SECONDARY OUTCOMES:
A secondary outcome is the staging power of PET/MRI compared to preoperative A-US (Axillary Ultrasound) | At 12 months
  Study will focus on a subgroup of patients having one or two uncertain but no suspicious axillary nodes for which SNB is still indicated. Patient population will be divided into two cohorts: those with completely normal axillary lymph node at A-US and those with 1-2 axillary nodes with uncertain ultrasound features. These two groups will be analysed independently. The PET/MRI and A-US results will be compared to each other and ultimately to final pathology, calculating the concordance rate in terms of positive versus negative nodes and number of positive nodes detected by each method. The staging power of both preoperative exams will be evaluated by considering how many times the results from PET/MRI or A-US could have indicated the most appropriate axillary treatment according to pathological findings.
Correlation between PET/MRI parameters and breast cancer prognosis | 0 and 36 months
  Eventual associations between PET/MRI morphological and functional parameters with tumour prognostic features will be investigated.

CONTACTS AND LOCATIONS:
Overall Officials: ORESTE D GENTILINI, MD, Principal Investigator — Director Breast Unit
Locations (1):
- Oreste Davide Gentilini, Milan, MI, Italy

REFERENCES:
- [Background] Gentilini O, Veronesi U. Staging the Axilla in Early Breast Cancer: Will Imaging Replace Surgery? JAMA Oncol. 2015 Nov;1(8):1031-2. doi: 10.1001/jamaoncol.2015.2337. No abstract available. PMID 26291922
- [Background] Pilewskie M, Jochelson M, Gooch JC, Patil S, Stempel M, Morrow M. Is Preoperative Axillary Imaging Beneficial in Identifying Clinically Node-Negative Patients Requiring Axillary Lymph Node Dissection? J Am Coll Surg. 2016 Feb;222(2):138-45. doi: 10.1016/j.jamcollsurg.2015.11.013. Epub 2015 Nov 25. PMID 26711795
- [Background] Heusch P, Nensa F, Schaarschmidt B, Sivanesapillai R, Beiderwellen K, Gomez B, Kohler J, Reis H, Ruhlmann V, Buchbender C. Diagnostic accuracy of whole-body PET/MRI and whole-body PET/CT for TNM staging in oncology. Eur J Nucl Med Mol Imaging. 2015 Jan;42(1):42-8. doi: 10.1007/s00259-014-2885-5. Epub 2014 Aug 12. PMID 25112399
- [Background] Stadnik TW, Everaert H, Makkat S, Sacre R, Lamote J, Bourgain C. Breast imaging. Preoperative breast cancer staging: comparison of USPIO-enhanced MR imaging and 18F-fluorodeoxyglucose (FDC) positron emission tomography (PET) imaging for axillary lymph node staging--initial findings. Eur Radiol. 2006 Oct;16(10):2153-60. doi: 10.1007/s00330-006-0276-4. Epub 2006 May 3. PMID 16670863
- [Background] Taneja S, Jena A, Goel R, Sarin R, Kaul S. Simultaneous whole-body (1)(8)F-FDG PET-MRI in primary staging of breast cancer: a pilot study. Eur J Radiol. 2014 Dec;83(12):2231-2239. doi: 10.1016/j.ejrad.2014.09.008. Epub 2014 Sep 28. PMID 25282709
- [Background] Melsaether AN, Raad RA, Pujara AC, Ponzo FD, Pysarenko KM, Jhaveri K, Babb JS, Sigmund EE, Kim SG, Moy LA. Comparison of Whole-Body (18)F FDG PET/MR Imaging and Whole-Body (18)F FDG PET/CT in Terms of Lesion Detection and Radiation Dose in Patients with Breast Cancer. Radiology. 2016 Oct;281(1):193-202. doi: 10.1148/radiol.2016151155. Epub 2016 Mar 29. PMID 27023002
- [Background] Veronesi U, De Cicco C, Galimberti VE, Fernandez JR, Rotmensz N, Viale G, Spano G, Luini A, Intra M, Veronesi P, Berrettini A, Paganelli G. A comparative study on the value of FDG-PET and sentinel node biopsy to identify occult axillary metastases. Ann Oncol. 2007 Mar;18(3):473-8. doi: 10.1093/annonc/mdl425. Epub 2006 Dec 12. PMID 17164229
- [Background] van Nijnatten TJA, Goorts B, Voo S, de Boer M, Kooreman LFS, Heuts EM, Wildberger JE, Mottaghy FM, Lobbes MBI, Smidt ML. Added value of dedicated axillary hybrid 18F-FDG PET/MRI for improved axillary nodal staging in clinically node-positive breast cancer patients: a feasibility study. Eur J Nucl Med Mol Imaging. 2018 Feb;45(2):179-186. doi: 10.1007/s00259-017-3823-0. Epub 2017 Sep 14. PMID 28905091
- [Derived] Di Micco R, Botteri E, Canevari C, Gallivanone F, Antunovic L, Scifo P, Neri I, Gelardi F, Magnani P, Losio C, Venturini E, Della Vecchia G, Ferrarese G, Rotmensz N, Zuber V, Baleri S, Cisternino G, Calabretto F, Corona SP, Rampa M, Pitoni L, Scaduto V, Morgante MM, Critelli A, Sassi I, Bianchini G, Panizza P, Chiti A, Gentilini OD. [18F]FDG PET/MRI vs sentinel node biopsy for axillary staging of early breast cancer patients. A prospective single-arm trial. Eur J Cancer. 2025 Jun 25;224:115519. doi: 10.1016/j.ejca.2025.115519. Epub 2025 May 24. PMID 40449294